CLINICAL TRIAL: NCT00208390
Title: Prospective, Uncontrolled, Multi-Centre, Post-Marketing Surveillance Study to Evaluate the Long-Term Performance of Summit Tapered Hip in Cementless Total Hip Arthroplasty
Brief Title: A Multi-centre Study to Assess the Long-term Performance of the Summit™ Hip in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed after the 5 year end-point was reached after a review of the status further to a request from the investigators to discontinue participation.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT01/25
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cementless
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Summit Tapered Hip System (Other): A cementless, tapered femoral component for use in total hip replacement
  Interventions: Device: Summit Tapered Hip System

INTERVENTIONS:
Device: Summit Tapered Hip System — A cementless, tapered femoral component for use in total hip replacement

SUMMARY:
The purpose of this study is to monitor the performance of the Summit™ hip in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 18 and 70 years (inclusive).

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects who require primary total hip replacement and are considered suitable for a cementless femoral stem.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Subjects who have previously undergone a hemi-arthroplasty or total hip arthroplasty.

iii) Women who are pregnant.

iv) Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.

v) Subjects who have participated in a clinical study with an investigational product in the last 12 months.

vi) Subjects who are currently involved in any injury litigation claims.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2003-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship calculated at the five-year time point | 5yrs post-surgery

SECONDARY OUTCOMES:
Kaplan-Meier survivorship calculations | Annually
Harris Hip score | 6mths, 1yr, 2yrs, 3yrs, 5yrs, 7yrs, 10yrs and 15yrs post-surgery
Oxford score | 6mths and Annually post-surgery
UCLA activity rating | 6mths and Annually post-surgery
Thigh pain analysis | 6mths and Annually post-surgery
Radiological analysis | pre-discharge, 6mths, 1yr, 2yrs, 3yrs, 5yrs, 7yrs, 10yrs and 15yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (5):
- 2. Ruijin Hospital, Shanghai, China
- 3. The University of Hong Kong at Queen Mary Hospital, Pokfulam, Hong Kong
- 1. Ospedale Riuniti Di Bergamo, Bergamo, Italy
- 5. Middlemore Hospital, Auckland, New Zealand
- 4. Yonsei University College of Medicine, Seoul, South Korea